CLINICAL TRIAL: NCT04111965
Title: Phase I-II Clinical Trial to Compare the Safety and Efficacy of Nanodrop® Against Systane® Balance in the Treatment of Dry Eye Patients
Brief Title: Clinical Trial to Compare the Safety and Efficacy of Nanodrop®
Acronym: PRO-176/I
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH176-1218/I-II
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Dry Eye
Keywords: Dry eye; propylene glycol
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Propylene Glycol

STUDY DESIGN:
Intervention Model Description: Phase I-II clinical trial, comparative, non-inferiority with active control, double blind with randomisation. Safety analysis when completing the visits of the first 12 subjects
Who Masked: Participant, Investigator
Masking Description: Masking will be done through the primary and secondary packaging.
  They will be identified by means of identical tags. Which, in compliance with current and applicable regulations, must contain at least:
  * Name, address and telephone number of the sponsor.
  * Pharmaceutical form and route of administration.
  * Lot Number.
  * Legend "Exclusively for clinical studies"
  * Date of Expiry.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nanodrop® (PRO-176) (Experimental): - Nanodrop®. 0.6% propylene glycol. Ophthalmic emulsion Laboratorios Sophia, S.A. from C.V. Route of administration: Ophthalmic.
  Interventions: Drug: Nanodrop®
- Systane® Balance (Active Comparator): * Systane® Balance. 0.6% propylene glycol. Ophthalmic emulsion Alcon Laboratories, Inc.
  * Route of administration: Ophthalmic.
  Interventions: Drug: Systane Balance

INTERVENTIONS:
Drug: Nanodrop® — minimum to meet 1 drop 4 times a day, both eyes
  Other Names: PRO-176; Propylene glycol 0.6%
  Arms: Nanodrop® (PRO-176)
Drug: Systane Balance — minimum to meet 1 drop 4 times a day, both eyes
  Other Names: Propylene glycol 0.6%
  Arms: Systane® Balance

SUMMARY:
Study design:

Phase I-II clinical trial, comparative, non-inferiority with active control, parallel groups, double blind with randomisation. Safety analysis when completing the visits of the first 12 subjects of the Nanodrop® group, if there are less than 20% of unexpected Events (EA), related to the research product, recruitment is continued until the sample is completed for efficacy analysis

objectives Security: Evaluate the safety of the ophthalmic application of Nanodrop® by quantifying the incidence of unexpected Adverse Events (EA) related to the research product (PI).

Effectiveness: Demonstrate the non-inferiority of Nanodrop® compared to Systane® Balance, in the efficacy of the treatment of patients with dry eye, by means of the Ocular Surface Disease Index (OSDI).

Hypothesis

Security:

H0 = Nanodrop® is safe in its ophthalmic application as it presents an incidence of unexpected adverse events related to the research drug, less than 20% of the population of Nanodrop® safety group.

H1 = Nanodrop® is not safe in its ophthalmic application, as it presents an incidence of unexpected adverse events related to the research drug, exceeding 20% of the population of Nanodrop® safety group.

Effectiveness:

H0 = Nanodrop® is lower than Systane® Balance by more than 5 points in the OSDI test score.

H1 = Nanodrop® is lower than Systane® Balance by 5 points or less in the OSDI test score.

Number of subjects: n = 126 evaluable subjects 63 evaluable subjects per group (both eyes).

Main inclusion criteria: Dry eye diagnosis

Duration of intervention treatment: 28 days Approximate duration of the subject in the study: 35 days

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to voluntarily grant your signed informed consent
* Power and willingness to comply with scheduled visits treatment plan and other study procedures
* Be willing to modify the activities of your lifestyle.
* Be of legal age
* Women of reproductive age should ensure continuation (initiated ≥ 30 days prior to the signing of the Informed Consent Form or ICF) of using a hormonal contraceptive method or intrauterine device (IUD) during the study period
* Present a dry eye diagnosis, defined by:

OSDI ≥ 13 points plus one of the following:

* Corneal staining with more than 5 sites
* Conjunctival staining with more than 9 sites
* Breakup Time of lacrimal film (BUT) <10 seconds:

Exclusion Criteria:

* In the case of women: being pregnant, breastfeeding or planning to get pregnant within the study period.
* Have participated in another clinical research study ≤ 30 days before the scrutiny visit.
* Having previously participated in this study.
* Present a Better Corrected Visual Acuity (MAVC) of 20/200 or worse in one of the eyes.
* Present an added ophthalmological diagnosis of:

Allergic, viral or bacterial conjunctivitis. Anterior blepharitis. Demodex. Eye parasitic infections. Unresolved eye trauma. Healing diseases of the ocular surface. Corneal or conjunctival ulcers. Filamentous keratitis. Neurotrophic keratitis. Bullous keratopathy. Neoplastic diseases on the ocular surface or annexes. Diseases with fibrovascular proliferations on the conjunctival and / or corneal surface.

Diseases in the retina and / or posterior segment that require treatment or threaten the visual prognosis.

Glaucoma

* Have a management of your dry eye that requires the implementation of stage 2 treatments of the recommendations in the treatment and management by stages for the dry eye disease from the Dry Eye Workshop II of The Tear Film and Ocular Surface Society (DEWS II, TFOS).
* Have a history of drug addiction or current drug dependence or within the last two years prior to the signing of the Informed Consent Form.
* Have a history of ocular surgical procedure within the last 3 months prior to the signing of the Informed Consent Form.
* Be a user of soft or hard contact lenses. You can enter if you can suspend your use during the study, you must turn 15 days without using the contact lens before inclusion.
* Having another medical condition, acute or chronic, that at the discretion of the researcher could increase the risk associated with participation in the study or administration of the product under investigation, or that could interfere with the interpretation of the results of the study.
* Present known hypersensitivity to the components of the products under investigation.
* Be or have an immediate family member (for example: spouse, parent / legal guardian, brother or child) who is an employee of the research site or the sponsor, and who participates directly in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Baiza Durán, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (6):
- Mexico (6):
  - Catarata y Glaucoma de Occidente, Guadalajara, Jalisco
  - Clínica de Investigación en Reumatología y Obesidad S.C., Guadalajara, Jalisco
  - Jose Navarro Partida, Guadalajara, Jalisco
  - Health Pharma Professional Research S.A. de C.V., Mexico City, Mexico City
  - Asociación para Evitar la Ceguera en México, I.A.P., Mexico City, Mexico City
  - Centro Potosino de Investigación Médica SC, San Luis Potosí City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baiza-Duran LM, Munoz-Villegas P, Sanchez-Rios A, Olvera-Montano O. Efficacy and Safety of an Ophthalmic DMPC-Based Nanoemulsion in Patients with Dry Eye Disease: A Phase I/II Randomized Clinical Trial. J Ophthalmol. 2023 Apr 10;2023:1431473. doi: 10.1155/2023/1431473. eCollection 2023. PMID 37077305

RESULTS

PARTICIPANT FLOW:
Groups:
- Systane® Balance: * Systane® Balance. 0.6% propylene glycol. Ophthalmic emulsion Alcon Laboratories, Inc.
  * Route of administration: Ophthalmic.
  Systane Balance: minimum to meet 1 drop 4 times a day, both eyes
Period: Overall Study
Arm/Group | Nanodrop® (PRO-176) | Systane® Balance
Started | 63 | 63
Completed | 56 | 59
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Population: The manifested adverse events during the conduction of this trial were obtained during trial visits and reported in the electronic CRF, where the clinical team of the center included the information from source documents. These were previously checked by the monitor team, pharmacovigilance specialist, and the medical specialist part of the sponsor's crew to verify concordance with what was stipulated in the protocol.
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Nanodrop® (PRO-176) | Systane® Balance | Total
Number analyzed (Participants) | 63 | 63 | 126
Number analyzed (Eyes) | 126 | 126 | 252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 57 | 110
  >=65 years | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (17.4) | 44.6 (15.4) | 46.18 (16.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 40 | 87
  Male | 16 | 23 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 63 | 63 | 126
Intraocular Pressure (IOP) [Mean (Standard Deviation); unit: mmhg] | 13.8 (3.1) | 12.7 (2.5) | 13.20 (3.41)

OUTCOME MEASURES:

1. Primary Outcome: Ocular Surface Disease Index (OSDI)
Description: OSDI is a questionnaire designed to measure eye surface irritation with Rasch analysis to produce estimates on a linear interval scale.. The OSDI score ranges from 0 to 100, with higher scores indicating greater severity of symptoms. A score of 0 represents no symptoms, while 100 represents the most severe symptoms.
Time Frame: will be evaluated at the end of the treatment (day 29, final visit)
Population: The evaluated population for this outcome measure was the PP population (subjects who finished the study without presenting any mayor deviations to protocol)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nanodrop® (PRO-176) | Systane® Balance
Number analyzed (Participants) | 54 | 59
score on a scale | 48.9 (19.2) | 50.3 (18.3)

2. Primary Outcome: Percentage of Unexpected Adverse Events (AE) Related to the Research Product
Description: the adverse events will be evaluated with a scale of Present / Absent, it is a nominal variable, the normal value is absent
Time Frame: during the 29 days of evaluation, including the safety call
Population: This outcome measure considered the Intention-To-Treat (ITT) population, all participants who were randomized and exposed to treatment, regardless of whether they adhered to the study protocol.
Measure: Number; unit: percentage of unexpected related AE
Arm/Group | Nanodrop® (PRO-176) | Systane® Balance
Number analyzed (Participants) | 63 | 63
percentage of unexpected related AE | 23.0 | 17.5

3. Secondary Outcome: Visual Acuity (VA)
Description: Visual acuity (VA) is a test of visual function. It will be evaluated with the Snellen chart. The Snellen chart is the standard tool used to evaluate visual acuity. It was located in a place with adequate lighting, natural or artificial and at a distance of 3 meters from the subject to be evaluated. The contralateral eye to which it will be evaluated is covered, then the examiner detects until the line can clearly see the letters given he or she a score, the normal score for a VA is 20/20.This score can be expressed in fraction (i.e. 20/20) decimal (i.e. 1.0), or LogMAR (i.e. 0) formats. In this study, VA is expressed in decimal format. In decimal format, a lower number is a worse outcome.
Time Frame: will be evaluated at the end of the treatment (day 29, final visit)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: decimal score (Snellen Chart)
Arm/Group | Nanodrop® (PRO-176) | Systane® Balance
Number analyzed (Participants) | 54 | 59
decimal score (Snellen Chart) | 0.89 (0.18) | 0.90 (0.19)

4. Secondary Outcome: Epithelial Defects (ED) Fluorescein Stain
Description: The epithelial defects will be evaluated by fluorescein, it is a discrete variable that will be realized by direct observation, It will be qualified according to the Eye Staining Rating (CTO) of the International Alliance of Clinical Collaboration of Sjögren (SICCA).According to the CTO, grade 0 corresponds to the absence of dotted epithelial erosions (EEP); Grade 1 is defined as the presence of 1-5 EEP; Grade 2 corresponds to 6-30 EEP; and> 30 EEP will be classified as grade 3. Additionally a qualification point will be added if: 1) EEP is presented in the central portion of the cornea with a diameter of 4mm; 2) filaments are observed and 3) confluent staining patches are observed, including linear stains. A greater score is a worse outcome.
Time Frame: will be evaluated at the end of the treatment (day 29, final visit)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Nanodrop® (PRO-176) | Systane® Balance
Number analyzed (Participants) | 54 | 59
Number analyzed (Eyes) | 108 | 118
score on a scale | 0.91 (0.92) | 0.93 (1.14)

5. Secondary Outcome: Epithelial Defects (ED) Green Lissamine
Description: The epithelial defects will be evaluated by green lissamine, it is a discrete variable that will be realized by direct observation, It will be qualified according to the Eye Staining Rating (CTO) of the International Alliance of Clinical Collaboration of Sjögren (SICCA). In the CTO, grade 0 is defined as the presence of 0 to 9 lissamine green staining points in the interpalpebral bulbar conjunctiva (qualifying the temporal and nasal portion separately); grade 1 is defined by the presence of 10 to 32 points; grade 2 by 33 to 100; and grade 3 for> 100 points. Due to the difficulty of counting individual points in a moving eye, any area ≥ 4mm2 of confluent points is considered> 100 points. A higher score is a worse outcome.
Time Frame: will be evaluated at the end of the treatment (day 29, final visit)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Nanodrop® (PRO-176) | Systane® Balance
Number analyzed (Participants) | 54 | 59
Number analyzed (Eyes) | 108 | 118
score on a scale | 0.83 (0.69) | 0.85 (0.78)

6. Secondary Outcome: Incidence of Expected Adverse Events
Description: as for outcome 2
Time Frame: will be evaluated at the end of the treatment (day 29, final visit)
Population: as for outcome 2
Measure: Number; unit: percentage of adverse events per group
Arm/Group | Nanodrop® (PRO-176) | Systane® Balance
Number analyzed (Participants) | 63 | 63
percentage of adverse events per group | 77 | 82.5

7. Secondary Outcome: Tear Breakup Time (TBUT)
Description: brake up time of the tear film One of the first aspects of the tear film that changes when there is an alteration to the ocular surface is its stability. In general, if the corneal or conjunctival surface is damaged, it is unlikely that a stable tear film can be maintained.
  The most common method to evaluate tear film stability is the evaluation of TBUT with fluorescein. Once the fluorescein is instilled, with the cobalt blue filter the patient is asked not to blink after having blinked 1 to 2 times. The colored precorneal fluorescein layer will change to less fluorescent or non-fluorescent regions. The time that elapses from the last blink to the appearance of these regions is the TBUT. It will be reported in seconds.
Time Frame: will be evaluated at the end of the treatment (day 29, final visit)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: reported in seconds
Arm/Group | Nanodrop® (PRO-176) | Systane® Balance
Number analyzed (Participants) | 54 | 59
reported in seconds | 2.28 (2.9) | 2.02 (2.9)

ADVERSE EVENTS:
Time Frame: Time frame will be evaluated from day 1 (basal visit) to the final visit day 28 (±1 days).
Description: The manifested adverse events during the conduction of this trial were obtained during trial visits and reported in the electronic CRF, where the clinical team of the center included the information from source documents. These were previously checked by the sponsor's monitor team, the pharmacovigilance specialist, and the medical specialist to verify adherence to procedures stipulated in the protocol.
Arm/Group | Nanodrop® (PRO-176) | Systane® Balance
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 1/63
Other Adverse Events (participants affected / at risk) | 54/63 | 47/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nanodrop® (PRO-176) (N=63) | Systane® Balance (N=63)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nanodrop® (PRO-176) (N=63) | Systane® Balance (N=63)
Burning sensation (Eye disorders) | 37 | 23
Irritation in the area of instillation (Eye disorders) | 5 | 3
sensation of ocular pain (Eye disorders) | 3 | 4
pruritus (Eye disorders) | 11 | 13
blurred vision (Eye disorders) | 4 | 11
ineffective drug (Product Issues) | 13 | 16
conjunctival hyperemia (Eye disorders) | 8 | 8
tearing (Eye disorders) | 1 | 5
headache (Nervous system disorders) | 7 | 1
asthenopia (Eye disorders) | 2 | 2
corneal lesion (Eye disorders) | 1 | 0
conjunctivitis (Eye disorders) | 4 | 2
epistaxis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT04111965/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT04111965/SAP_001.pdf